CLINICAL TRIAL: NCT03081611
Title: RAM Cannula for Delivering Nasal Intermittent Positive Pressure Ventilation (NIPPV) in Preterm Infants: Non Inferiority Randomized Control Trial
Brief Title: RAM Cannula VS Short Nasal Prongs for Delivering NIPPV in Preterm Infants
Acronym: RAMCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ori Hochwald , MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAMCAN
Record Dates: First submitted 2017-03-12; First posted 2017-03-16 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Respiratory Distress Syndrome, Newborn; Noninvasive Ventilation; Infant, Premature; Intubation, Intratracheal
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth

STUDY DESIGN:
Intervention Model Description: Non Inferiority Randomized Control Trial
Masking Description: Not possible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ram cannula (Experimental): NIPPV VIA Ram cannula
  Interventions: Device: Ram cannula
- Short nasal prongs (Active Comparator): NIPPV VIA short nasal prongs
  Interventions: Device: Short nasal prongs

INTERVENTIONS:
Device: Ram cannula — Ventilatory support for preterm infants using Ram cannula
  Arms: Ram cannula
Device: Short nasal prongs — Ventilatory support for preterm infants using short nasal prongs
  Arms: Short nasal prongs

SUMMARY:
Randomized control trial, Ram cannula VS short nasal prongs for delivering Non Invasive Positive Pressure Ventilation (NIPPV) for preterm infants

DETAILED DESCRIPTION:
Randomized control trial comparing Ram cannula to the regular, more investigated short nasal prongs for delivering Non Invasive Positive Pressure Ventilation (NIPPV) for preterm infants with respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 24-33.6
* Physician decision on the need for non invasive ventilation
* parental consent

Exclusion Criteria:

* Pneumothorax before recruitment
* Significant congenital heart disease or chromosomal disorder

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
intubation | 72 hours
  The need for intubation

SECONDARY OUTCOMES:
nasal trauma | during NIPPV procedure
  nasal trauma

CONTACTS AND LOCATIONS:
Overall Officials: Ori Hochwald, MD, Principal Investigator — NICU, Rambam Medical Center, Haifa, Israel
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hochwald O, Riskin A, Borenstein-Levin L, Shoris I, Dinur GP, Said W, Jubran H, Littner Y, Haddad J, Mor M, Timstut F, Bader D, Kugelman A. Cannula With Long and Narrow Tubing vs Short Binasal Prongs for Noninvasive Ventilation in Preterm Infants: Noninferiority Randomized Clinical Trial. JAMA Pediatr. 2021 Jan 1;175(1):36-43. doi: 10.1001/jamapediatrics.2020.3579. PMID 33165539